CLINICAL TRIAL: NCT05530824
Title: Satisfaction Survey for the Outpatient Unit Dedicated to Post-cancer Treatment
Acronym: BAC
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: BAC
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Ambulatory
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The care pathway for breast cancer is complex, punctuated by consultations, complementary examinations and treatments. Patients benefit from close medical and paramedical support. At the end of the treatment, the post-cancer phase begins and the surveillance begins. The National Cancer Institute's (INCa) ten-year cancer control strategy for 2021-2030 defines in its second axis the objective of limiting the after-effects and improving the quality of life of cancer patients. Indeed, ensuring rapid access to functional rehabilitation and post-treatment reconstruction, and setting up personalized and graduated follow-up between the city and the hospital, are crucial. Better information for patients on the post-cancer period is a way for them to acquire greater autonomy, to enable them to take an active role in it and to approach it with greater serenity.

The Paris Saint-Joseph Hospital Group (GHPSJ) has therefore created an outpatient medical unit (UMAb) dedicated to post-cancer treatment in July 2021. It is offered to all patients who have had localized breast cancer and have received curative treatment. Each patient, 3-4 months after the end of treatment (surgery and/or chemotherapy and/or radiotherapy), will benefit from a half-day session including 3 consultations: medical, nursing and physiotherapy. The medical consultation allows for additional information if there are any questions about the care received, a clinical examination, reassessment of the tolerance of adjuvant hormone therapy if it is indicated, and delivery of the personalized post-cancer program (PPAC). The nursing consultation is conducted by a person certified in therapeutic patient education. Numerous items are discussed, with the aim of identifying personal difficulties (financial, family or work-related, for example) that may hinder post-cancer rehabilitation, detecting specific support care needs and promoting post-cancer health (encouraging normal weight, smoking cessation, recommended nutritional factors and physical activity). Finally, the physical therapy consultation consists of a joint, muscle and scar assessment to promote normal functionality and the implementation of recommended physical activity. Imaging examinations (cardiac ultrasound and/or mammography/ultrasound and/or bone densitometry) may be associated with the consultation.

As part of investigator's quality and continuous improvement approach, investigators would like to collect the opinions of patients who have benefited from the UMAb post breast cancer since its creation.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age is ≥ 18 years
* Patient who has participated in post-cancer UMAB for breast cancer
* French-speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of her data for this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient whose age is ≥ 18 years, who has participated in post-cancer UMAB for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Satisfaction reported by patients regarding the implementation of UMAb post breast cancer | Month 1
  This outcome corresponds to the number of satisfied patients who felt a benefit after participating in UMAb post breast cancer, using the satisfaction questionnaire.

SECONDARY OUTCOMES:
Improvement in the post-breast cancer AMU | Month 1
  This outcome corresponds to the patient expectations and areas for improvement in post-breast cancer UMAb.
Profile of patients with lower post-cancer UMAb scores to optimize their management, with specific measures | Monthe 1
  This outcome corresponds to the characteristics of patients with lower post-cancer UMAb scores (Scale: Very dissatisfied, Dissatisfied, Neutral, Satisfied, Very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Olivia NGUYEN, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] de Boer AG, Taskila T, Ojajarvi A, van Dijk FJ, Verbeek JH. Cancer survivors and unemployment: a meta-analysis and meta-regression. JAMA. 2009 Feb 18;301(7):753-62. doi: 10.1001/jama.2009.187. PMID 19224752
- [Background] Duijts SF, van Egmond MP, Spelten E, van Muijen P, Anema JR, van der Beek AJ. Physical and psychosocial problems in cancer survivors beyond return to work: a systematic review. Psychooncology. 2014 May;23(5):481-92. doi: 10.1002/pon.3467. Epub 2013 Dec 23. PMID 24375630
- [Background] Spei ME, Samoli E, Bravi F, La Vecchia C, Bamia C, Benetou V. Physical activity in breast cancer survivors: A systematic review and meta-analysis on overall and breast cancer survival. Breast. 2019 Apr;44:144-152. doi: 10.1016/j.breast.2019.02.001. Epub 2019 Feb 12. PMID 30780085